CLINICAL TRIAL: NCT00321542
Title: Assessment of the Additive Value of Multislice Computed Tomographic Angiography of the Coronary Arteries in the Prediction of Acute Cardiac Events in Asymptomatic Individuals With Type II Diabetes Mellitus
Brief Title: Coronary CT Angiography in Asymptomatic Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Other Study IDs: CT-DM
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus
Keywords: Computed tomography; Diabetes mellitus; Coronary atherosclerosis; Non-invasive imaging
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Imaging study, No intervention — Imaging with coronary computed tomographic angiography
  Other Names: Philips Brilliance 64 computed tomography scanner

SUMMARY:
The study aims to examine if non-invasive imaging of the coronary arteries by CT angiography using an intra-venous injection of X-ray contrast medium in asymptomatic patients with adult onset diabetes mellitus can predict the risk of developing coronary heart disease.

DETAILED DESCRIPTION:
Patients having diabetes mellitus are at increased risk for the development of coronary heart disease. Available tests do not accurately predict which diabetic patients are at greatest risk of suffering from a coronary event. The recent development of coronary CT angiography allows non-invasive imaging of both coronary narrowing and of disease (atheroma) in the coronary arterial wall at an earlier stage of the disease before the development of coronary arterial narrowing.

In this study we will collect all the readily available patient medical data relating to diabetes and its complications and other coronary artery disease risk factors. In addition patients will be referred for exercise stress testing and for eye examinations. The coronary CT angiogram will be carefully examined for early signs of coronary artery disease. In the event of a finding on the CT scan requiring medical therapy this will be communicated to the patient and his treating physician. In the event of a finding on the stress test or CT scan requiring further medical work-up the patient will be referred to the cardiology clinic.

In general patients will be followed in the regular diabetic clinic and by their family practitioners.

In the event of any acute symptoms over the next few years possibly related to heart disease and requiring emergency room examination patients will be requested to report to the emergency room at the hospital at which the CT study was performed whenever possible.In such an event a repeat CT scan will be performed to examine if any new findings are present. In the event of any new complaints requiring referral to an out of hospital clinic patients will be referred for further assessment to the cardiology clinic and a repeat CT scan may be performed if deemed relevant.

Outcomes of all patients will be examined at 2 years or later using computerized databases. Patients undergoing hospitalization during the follow up period of at least 2-3 years will be contacted by the study staff to obtain further details of the event and hospital findings .

An analysis wil be performed of the value of CT angiography in relation to the traditional risk factors and other available medical data in the prediction of later coronary heart disease and other vascular events.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus
* No symptoms of coronary heart disease
* At least one additional risk factor for coronary artery disease

Exclusion Criteria:

* Known coronary artery disease
* Kidney failure if more than mild
* Allergy to iodinated X-ray contrast media
* Chronic atrial fibrillation

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabtes mellitus, age 55-74 yrs, no known coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2006-09; Primary Completion 2015-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Death or acute myocardial infarction | 7 years

SECONDARY OUTCOMES:
Composite of the primary outcome and the onset of new symptoms of coronary artery disease with proven myocardial ischemia (supported by treadmill, nuclear scan or stress echo findings) or the need for a revascularization procedure. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: David A Halon, MB ChB, FACC, Study Director — Lady Davis Carmel Medical Center
Locations (1):
- Lady Davis Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Scognamiglio R, Negut C, Ramondo A, Tiengo A, Avogaro A. Detection of coronary artery disease in asymptomatic patients with type 2 diabetes mellitus. J Am Coll Cardiol. 2006 Jan 3;47(1):65-71. doi: 10.1016/j.jacc.2005.10.008. Epub 2005 Dec 9. PMID 16386666
- [Background] Leber AW, Knez A, von Ziegler F, Becker A, Nikolaou K, Paul S, Wintersperger B, Reiser M, Becker CR, Steinbeck G, Boekstegers P. Quantification of obstructive and nonobstructive coronary lesions by 64-slice computed tomography: a comparative study with quantitative coronary angiography and intravascular ultrasound. J Am Coll Cardiol. 2005 Jul 5;46(1):147-54. doi: 10.1016/j.jacc.2005.03.071. PMID 15992649
- [Derived] Halon DA, Dobrecky-Mery I, Gaspar T, Azencot M, Yaniv N, Peled N, Lewis BS. Pulse pressure and coronary atherosclerosis in asymptomatic type 2 diabetes mellitus: a 64 channel cardiac computed tomography analysis. Int J Cardiol. 2010 Aug 6;143(1):63-71. doi: 10.1016/j.ijcard.2009.01.066. Epub 2009 Feb 25. PMID 19246107